CLINICAL TRIAL: NCT05611697
Title: Laparoscopic Single Anastomosis Sleeve Ileal Bypass Versus Laparoscopic Sleeve Gastrectomy for Morbid Obesity: A Randomized Trial
Brief Title: Laparoscopic Single Anastomosis Sleeve Ileal Bypass Versus Laparoscopic Sleeve Gastrectomy for Morbid Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Torgeir Søvik, Principal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 319260
Record Dates: First submitted 2022-05-09; First posted 2022-11-10 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Obesity, Morbid
Keywords: procedure: sleeve gastrectomy; bariatric surgery; procedure: single anastomosis sleeve ileal bypass
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Intervention Model Description: Patients are randomized in a 1:1 ratio to sleeve gastrectomy or SASI. The randomization list will contain block sizes of 4 and 6 in random order, stratified by study center.
Who Masked: Participant
Masking Description: Patients are allocated to surgical treatment 2 weeks before surgery and blinded to treatment allocation until the first postoperative day.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single anastomosis sleeve ileal bypass (Experimental): A Single anastomosis sleeve ileal bypass procedure is performed.
  Interventions: Procedure: Single anastomosis sleeve ileal bypass
- Sleeve gastrectomy (Active Comparator): A sleeve gastrectomy procedure is performed.
  Interventions: Procedure: Sleeve gastrectomy

INTERVENTIONS:
Procedure: Single anastomosis sleeve ileal bypass — The abdominal cavity is entered directly (visual trocar) with or without the use of Verres needle. A 6-port set up and a liver retractor is utilized. A sleeve gastrectomy is performed as described below, but division of the stomach starts 6 cm proximal to the pylorus. The small bowel is measured 300cm from the ileocecal valve, with the small bowel stretched and markers placed on the graspers, and connected to the antrum of the stomach with a 45mm stapler. The anastomosis is positioned slightly ventral on the antrum. A 12 mm port positioned left to the midline is used for introduction of the stapler, which is directed distally from the patient's left to right side. 3.0 cm of 45 mm stapler is used the anastomosis; completed with a 2-0 PDS running suture. The biliopancreatic limb is anchored to the sleeve 4 cm proximal to the anastomosis (non-resorbable V-loc 3-0). Fascia defect is closed for the port where the specimen is extracted. The mesenteric defect is not closed.
  Other Names: SASI
  Arms: Single anastomosis sleeve ileal bypass
Procedure: Sleeve gastrectomy — In the laparoscopic sleeve gastrectomy, the abdominal cavity is entered directly with a visual trocar with or without the use of Verres needle. The set up includes a total of 5 ports. The Natanson liver retractor is utilized. The greater omentum is separated from the major side of the stomach from the pylorus to the angle of His. The left crus is visualized and the hiatus is inspected for the presence of hernia. A 36 French bougie is introduced and the stomach is divided along this from 4-5cm proximal to the pylorus to 1cm lateral to the angle of His using two purple cartridges (Medtronic Tri-Staple™ technology) followed by beige 60mm cartridges to the angle of His, 1 cm lateral to the esophagus. The sleeve is tested for leaks with instillation of 50ml methylene blue in the tube. The fascia defect is closed with suture for the port site where the specimen is extracted.
  Arms: Sleeve gastrectomy

SUMMARY:
This study will compare two bariatric surgical interventions in terms of weight loss, gastroesophageal reflux, and effects on obesity-related comorbid conditions in morbidly obese patients.

DETAILED DESCRIPTION:
Sleeve gastrectomy is an established therapeutic option for morbidly obese patients without preexisting gastroesophageal reflux disease. The novel single anastomosis sleeve ileal bypass (SASI) procedure is already introduced in Norway at a private high-volume bariatric hospital. The purpose of this study is to evaluate the effects of SASI in comparison to an established bariatric procedure, i.e. sleeve gastrectomy. The primary end point is 2-year changes in BMI after sleeve gastrectomy and SASI.

ELIGIBILITY:
Inclusion Criteria:

1. Morbid obesity at referral for bariatric surgery (i.e. a body-mass index [BMI] of ≥35 kg/m2 with obesity-related comorbid conditions or ≥40 kg/m2 with or without such comorbidities).
2. Age 20-60 years.
3. Previous failed attempts of weight loss.
4. Norwegian speaking patients.

Exclusion Criteria:

1. BMI ≥55 kg/m2.
2. A history of major abdominal or bariatric surgery (excluding appendectomy, cholecystectomy, and sectio).
3. Established disabling cardiopulmonary disease, ongoing treatment for cancer, long-term steroid use, and conditions believed to be associated with poor adherence after surgery.
4. Previous or current gastroesophageal reflux symptoms with daily use of antireflux medication. Patients are also excluded if preoperative manometry identifies a hiatal hernia (≥4cm in axial length) or if preoperative upper endoscopy identifies esophagitis grade C or D (LA classification), peptic stricture, Barrett's esophagus, or esophageal carcinoma.
5. Achalasia
6. Pregnancy.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-02-17 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Changes in body-mass index (BMI) | 2 year
  Weight in kilograms divided by the square of the height in meters after sleeve gastrectomy and SASI.

SECONDARY OUTCOMES:
Change in prevalence of esophagitis. | 2 year
  Changes in the prevalence of esophagitis as evaluated by upper endoscopy.
Change in prevalence of gastroesophageal reflux disease. | 2 year
  Changes in the prevalence of gastroesophageal reflux disease as evaluated by 24-hour pH measurements.
Complications | 6 weeks (100 days for deaths), 2 year, 5 year
  Complications during surgery, postoperative complications (within 6 weeks [100 days for deaths]) as defined by the Accordion severity grading system and long-term complications.
Obesity-related comorbid conditions. | 2 year, 5 year
  Changes in obesity-related comorbid conditions.
Vitamin concentrations | 2 year, 5 year
  Changes in vitamin levels (A, B1, B6, B9, B12, C, D, K).
Health-related quality of life | 2 year, 5 year
  The RAND 36-Item Short Form Health Survery is a self-reporting questionnaire. Items are scored from 0 (lowest score) to 100 (highest possible score).
Obesity-related symptoms | 2 year, 5 year
  Obesity-related Problem scale
Gastrointestinal symptoms | 2 year, 5 year
  GSRS
Gastroesophageal reflux disease symptoms | 2 year, 5 year
  GERDq
Bowel habits | 2 year, 5 year
  Bowel habit questionnaire
Revisional surgery | 2 year, 5 year
  Revisional surgery rates in the two groups.
Long-term changes in BMI | 5 years
  BMI (weight in kilograms divided by the square of the height in meters) after sleeve gastrectomy and SASI.
Body composition | 2 years
  Changes in percentage fat mass and lean mass; percentage change in bone mineral density in lumbar spine (L1-L4), femoral neck, and total hip as assessed by DEXA scan.

CONTACTS AND LOCATIONS:
Overall Officials: Torgeir T Søvik, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (2):
- Norway (2):
  - The Morbid Obesity Center, Vestfold Hospital Trust, Tønsberg, Vestfold
  - Oslo University Hospital, Oslo

IPD SHARING:
Plan to Share IPD: No